CLINICAL TRIAL: NCT02888366
Title: A Prospective Validation Study of a Rapid Point-of-Care Breath Test for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Menssana Research, Inc. (Industry)
Collaborators: University of Southern California (Other); M.D. Anderson Cancer Center (Other); Hackensack Meridian Health (Other); St. Michael's Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: MR2016-03
Record Dates: First submitted 2016-08-22; First posted 2016-09-05 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; breath test; Menssana; Ancillary; Mammography; Rapid Point-of-care; Inflatable Bag
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Breath samples taken, no treatment given.

SUMMARY:
This is a multicenter, blinded prospective study of 2,000 women undergoing mammography for breast -related symptoms or signs. Breath tests will be performed in order to demonstrate that the outcome of mammography results combined with breast test results improves clinical sensitivity and specificity in a group that has an increased prior probability of cancer. Breath will be collected and analyzed with a rapid point-of-care instrument (BreathLink™) and also with a laboratory-based assay of samples collected into an inflatable bag (BreathBag™).

DETAILED DESCRIPTION:
Introduction

Clinical perspective on breath testing for breast cancer:

Breast cancer is the most commonly diagnosed cancer in women, in whom it is second only to lung cancer as a cause of cancer death. The National Cancer Institute estimated that more than 232,000 US women would be diagnosed with breast cancer in 2013 and nearly 40,000 would die of the disease.

Screening mammography and its limitations: In order to reduce the number of breast cancer deaths, many countries have established screening mammography programs to detect and treat early-stage disease. However, the impact of screening mammography on mortality has been questioned. Also, screening mammography is limited by its very low yield: a 2005 retrospective analysis reported that 510 US radiologists performed 2,289,132 screening mammograms and found 9,030 cancers i.e. only one cancer was found for every 253 mammograms. 99.6% of all screening mammograms were negative for cancer: they provided reassurance, but at a human cost of millions of women exposed to potentially hazardous radiation and discomfort, and a financial cost of several million dollars. Also, screening mammography may be associated with an increased risk of radiation-induced breast cancer, as well as with overdiagnosis and overtreatment. Many women decide not to take the test even when it is readily available, and screening mammography may be underutilized because of fear of pain and radiation exposure, ethnicity, poverty, and level of education.

Breath tests - a new diagnostic tool: Abnormal volatile organic compounds (VOCs) in breath have been identified in breast cancer. Breath VOC biomarkers have been reported in other disorders including bronchial asthma, lung cancer, active pulmonary tuberculosis, radiation exposure, and heart transplant rejection. The Food & Drug Administration (FDA) approved the nitric oxide breath test in bronchial asthma, the urea breath test for H. pylori, and Menssana Research's Heartsbreath test for heart transplant rejection under the Humanitarian Device Exemption regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18 years or over
2. Referred for mammography for a breast-related concern (e.g. breast mass, nipple discharge etc.)
3. Understands the study, and is willing to give written informed consent to participate
4. Approves collection of relevant additional data for clinical research record if and when it becomes available, including results of mammogram and any other imaging studies, biopsy results, TNM staging, and other relevant biomarker data e.g. status of BRCA1, BRCA2, HER2 and receptors (ER+ or ER-) and progesterone (PgR+ or PgR-)

Exclusion Criteria:

1. Known serious or potentially life-threatening disease (e.g. severe cardiac or infectious disease)
2. Previous history of treated breast cancer, or cancer of any other site, with the exception of basal cell carcinoma of skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2,000 women undergoing diagnostic mammography for breast-related symptoms or signs.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
A PROSPECTIVE VALIDATION STUDY OF A RAPID POINT-OF-CARE BREATH TEST FOR BREAST CANCER | 2 years
  Change in sensitivity and specificity of mammography for breast cancer when combined with results of breath test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Phillips, MD, Principal Investigator — Menssana Research, Inc.
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Hackensack Medical Center, Mountainside Hospital, Montclair, New Jersey
  - St. Michael's Medical Center, Newark, New Jersey
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided